CLINICAL TRIAL: NCT01412840
Title: Sterile Water Injections as a Complementary Method for Relieving Ureterolithiasis Pain- a Randomized Controlled Trial
Brief Title: Sterile Water Injections for Relieving Ureterolithiasis Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Skövde (Other)
Responsible Party: Principal Investigator, Lena B Martensson, Associate Professor, University of Skövde
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 787-08
Record Dates: First submitted 2010-11-24; First posted 2011-08-09 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Ureterolithiasis; Pain
Keywords: Ureterolithiasis; Pain; Complementary; RCT
MeSH Terms: conditions — Ureterolithiasis; Pain | interventions — Diclofenac; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard care and sterile water injections (Experimental): The patients in the intervention group will be given standard treatment, i.e. intramuscular injection of 50 mg diclofenac. Patients in this group will also be given four subcutaneous injections of 0.5 ml sterile water at the same segmental level, i. e. the area in which the patient reports the pain.
  Interventions: Other: Diclofenac and sterile water injections
- Standard care and isotonic saline (Placebo Comparator): The patients in this group will be given standard treatment, i.e. intramuscular injection of 50 mg diclofenac They will also be given four subcutaneous injections of isotonic saline at the same segmental level, i. e. the area in which the patient reports the pain.
  Interventions: Other: Diclofenac and isotonic saline
- Standard care (No Intervention): The patients in this group will be given standard treatment, i.e. intramuscular injection of 50 mg diclofenac.

INTERVENTIONS:
Other: Diclofenac and sterile water injections — The patients in the intervention group will be given standard treatment, i.e. intramuscular injection of 50 mg diclofenac. Patients in this group will also be given four subcutaneous injections of 0.5 ml sterile water at the same segmental level, i. e. the area in which the patient reports the pain.
  Arms: Standard care and sterile water injections
Other: Diclofenac and isotonic saline — The patients in this group will be given standard treatment, i.e. intramuscular injection of 50 mg diclofenac They will also be given four subcutaneous injections of isotonic saline at the same segmental level, i. e. the area in which the patient reports the pain.
  Arms: Standard care and isotonic saline

SUMMARY:
Ureterolithiasis pain is a severe condition for which it takes some 30 minutes for standard treatment to yield maximal pain relief, a period during which the patient suffers severe to intolerable pain. It would thus be valuable to further evaluate sterile water injection as a method for achieving rapid relief for this type of pain.

ELIGIBILITY:
Inclusion Criteria:

* Ureterolithiasis pain, acute onset,
* Requires pain relief,
* Standard treatment prescribed,
* Age 18-60,
* Ability to understand and follow instructions

Exclusion Criteria:

* Other administration of NSAID for analgesia 12 hours prior to intervention,
* Pregnancy with obstructed flow of urine

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in experience of pain | VAS before treatment and 1,5,10,15,20,30,60,90 and 12o minutes after treatment
  Measurement tool: Visual Analogue Scale (VAS)

SECONDARY OUTCOMES:
Requirement for additional pain relief | Reported in the protocol up to two hours after treatment
  The staff will reporter if any additional pain relief treatment have been used

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Bergh, PhD, Principal Investigator — University of Skövde
Locations (1):
- School of Life Sciences, University of Skövde, Skövde, Sweden